CLINICAL TRIAL: NCT01377272
Title: Spatial Epidemiology of HIV Infection
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Institute of Epidemiology, Institute of Epidemiology
Other Study IDs: 200808048R
Record Dates: First submitted 2008-10-22; First posted 2011-06-21 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-05

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: HIV/AIDS; spatial epidemiology; geographic information system; HIV-infection/Aids
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Data will be extracted from the National Taiwan University Hospital (NTUH) medical records database, geocoded according to the street address so that the case number, incidence, etc could be mapped. The spatial data would be used to detect the aggregation of HIV cases, existence of "hot spots" and then determine if they may merit further investigation or may have occurred by chance. The results from these GIS-based analyses would address local variations in HIV prevalence and transmission.

DETAILED DESCRIPTION:
The transmission routes of human immunodeficiency virus (HIV) are well known and many control programs focusing on risk groups and behavior have been undertaken. However, the risk factors of HIV transmission are not only at individual level (eg: demographic, behavior, and genetic risk factors), socioeconomic and environmental factors also take important roles. In Taiwan, few researches explored the spatial distribution of HIV infection. Studies in other countries observed a significant geographic variation in HIV infection. To understand the spatial pattern of HIV infection in depth, the present study aims to retrospectively investigate the epidemiological and geographic characteristics of HIV infection using the medical records database of National Taiwan University Hospital. A Geographic information system (GIS) and spatial statistics will be used to analyze the geographic patterns to determine whether spatial dispersion or clustering. There are two aims of this study. One is to investigate the epidemiology of HIV infection in Taipei City. The second is to analyze the spatial characterizes of HIV infection, including disease mapping, geographic correlation studies, and identifying the presence of HIV clusters and their potential spatial risk factors. In addition, we want to examine whether there are different distributions between different classificatory groups. Finally, we hope that our findings would give some direction for local health and policy planners to improve the HIV intervention and prevention strategies

ELIGIBILITY:
Inclusion Criteria:

* HIV/AIDS patients of NTUH

Exclusion Criteria:

* HIV/AIDS patient whose address cannot be geocoded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NTUH patients
Sampling Method: Non-Probability Sample
Enrollment: 1264 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Tai Fang, ph.D, Study Director — Institute of Epidemiology, National Taiwan University; Tzai-Hung Wen, ph.D, Study Director — Institute of Epidemiology, National Taiwan University; Ann-Chi Yang, bechelor, Principal Investigator — Institute of Epidemiology, National Taiwan University
Locations (1):
- Institute of Epidemiology, National Taiwan University, Taipei, Taiwan